CLINICAL TRIAL: NCT04936971
Title: Effect of the Introduction of mTor Inhibitors in the Activation of the Cytomegalovirus (CMV) -Specific Cellular Immune Response to Control Viral Replication in Kidney Transplant Patients
Brief Title: Introduction of mTor Inhibitors and the Activation of the Cytomegalovirus (CMV) -Specific Cellular Immune Response
Acronym: ACTIVA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Impossibility to perform tests (elispot) of the study due to change of location of laboratory
Sponsor: Edoardo Melilli (Other)
Responsible Party: Sponsor-Investigator, Edoardo Melilli, MD, PhD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACTIVA
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2021-06

CONDITIONS: Kidney Transplantation; Cytomegalovirus Infections
Keywords: Cytomegalovirus; kidney transplant; ELISPOT
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: Prospective, open label, randomized, two arms, paralel, compared to Standard of Care treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everolimus (Experimental): Kidney transplant induction with Rabbit Anti-Thymocyte globulin (rATG) as per local practice.
  Kidney transplant manteinance treatment with Tacrolimus (TAC) to achieve 4-6 ng/mL trough levels, Everolimus (EVL) to achieve 3-8 ng/mL trough levels and Corticosteroids (CS) as per local practice.
  Interventions: Other: no intervention
- Mycophenolate Mofetil (Active Comparator): Kidney transplant induction with Rabbit Anti-Thymocyte globulin (rATG) as per local practice.
  Kidney transplant manteinance treatment with Tacrolimus (TAC) to achieve 4-6 ng/mL trough levels, Mycofenolate Mofetil (MMF) 500mg/bid and Corticosteroids (CS) as per local practice.
  Interventions: Drug: Switch from Mycophenolate Mofetil to Everolimus manteinance treatment in Active Comparator Arm

INTERVENTIONS:
Drug: Switch from Mycophenolate Mofetil to Everolimus manteinance treatment in Active Comparator Arm — Switch from Mycophenolate Mofetil in Active comparator Arm if assymptomatic Cytomegalovirus viremia >1000-<5000 copies/mL observed
  Other Names: Switch to Certican
  Arms: Mycophenolate Mofetil
Other: no intervention — Manteinance of assigned Arm treatment even if assymptomatic Cytomegalovirus viremia >1000-<5000 copies/mL observed
  Arms: Everolimus

SUMMARY:
Kidney transplant patients under an immunosuppressive treatment based on anti-calcineurin and mycophenolate-mofetil and induction therapy with rATG who suffer from early systemic viral replication by the CMV virus could benefit from the introduction of an i-mTor drug. (everolimus) to replace mycophenolate mofetil. This conversion would be effective in slowing down and controlling viral expansion without the need to initiate any prophylactic anti-viral therapy thanks to the activation of the CMV-specific cellular effector response or to an antiviral effect of i-Mtor itself.

DETAILED DESCRIPTION:
Human cytomegalovirus (CMV) is the most common opportunistic pathogen in the first months after solid organ transplantation, being associated with an increased risk of acute and chronic graft rejection, graft loss and an increase in patient mortality.

The susceptibility to developing CMV infection is essentially determined by the host's immune status against the virus, with seronegative recipients (IgG-) receiving a graft from a seropositive donor (IgG +) (R- / D +) being the group with an especially high risk of developing CMV infection and disease after transplantation. In fact, without the administration of a preventive therapy for CMV, around 60-70% of this risk group will present viral infection (replication of copies of CMV in blood) and up to 30% will develop systemic disease (viral invasion of the tissue). However, the incidence of infection among R + / D + seropositive (IgG +) patients under treatment with induction with anti-IL2RA and the combination of mycophenolate mofetil (MPA) and anti-calcineurin drugs (CNI), can reach up to 40%, and up to 60% if induction therapies are administered with T-lymphocyte depletors with polyclonal antibodies (Thymoglobulin®, rATG) (6). All this suggests that the assessment of the immunological risk of developing post-transplant CMV infection is relatively poor and that the humoral response to the virus does not fully explain the patient's immunological susceptibility to the virus.

In this sense, it is well known that the subpopulation of CMV-specific memory / effector T cells plays a key role in the control of viral survival replication in general and of CMV in particular. While it has been reported that CD8 + cytotoxic T cells have the ability to activate against a wide range of immunogenic proteins of the CMV virus, it appears that high frequencies directed against the major CMV antigens such as those of immediate expression-1 (IE-1) and phosphoprotein 65 (pp65) play a critical role in the control of CMV viral replication. One of the most precise functional techniques to study the cellular memory immune response is the IFN-γ ELISPOT test, which allows knowing the antigen-specific response at the individual cellular level, thus providing high sensitivity and specificity. Along these lines, our group and others have shown how the monitoring of the CMV-specific cell response with the IFN-γ ELISPOT test, both before and after transplantation, is capable of identifying those patients with a high risk of developing infection by CMV, regardless of immunization status. In addition, data from a prospective, randomized clinical trial led by our group, evaluating the cellular response to CMV before transplantation using the IFN-γ ELISPOT test, have confirmed the high negative predictive power in identifying those patients with high risk of developing viral infection after transplantation, despite being serologically positive.

Mtor (mammalian target of rapamycin) inhibitors, everolimus and sirolimus, are a class of immunosuppressants commonly used in kidney transplantation both in the initial phase (de novo) and in the maintenance phase. In addition, today it is considered routine clinical practice in case of side effects mediated by CNI (tacrolimus or cyclosporine) or by antimetabolites (mycophenolate mofetil or mycophenolic acid) to replace the latter with iMtor (conversion to iMtor).

Interestingly, recently reported clinical studies have shown a significant decrease in the rate of both CMV infection and disease in patients treated with mTor inhibitors (i-mTOR) after kidney transplantation, both in combination with MPA. as in combination with CNI drugs. A recently published randomized clinical trial that included more than 2000 kidney transplant patients has reported that the incidence of CMV viral infection in the CNI plus everolimus group in the Serology D / R + / + group was 3.6% compared to 13.3% of the control group treated with CNI plus mycophenolate mofetil. (RR 0.27 - CI 0.19-0.38) This effect has been reported mainly among R + / D + patients, and even in those after receiving induction treatment with rATG.

Although the mechanism through which i-mTORs can inhibit and block viral replication after transplantation is unknown, it is suggested that it could be through their ability to directly inhibit proliferation on the virus, or well, through some of the immunomodulatory pleiotropic effects that they exert on the adaptive immune response. Along these lines, beyond its immunosuppressive capacity by inhibiting the lymphocyte proliferation signal

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years or older (and weigh more than 34Kg) and may be of both sexes and of any race.
2. Subjects will be seropositive for CMV virus and will receive a seropositive graft (CMV IgG D + / R +).
3. Subjects must be willing and able to give their written informed consent to the trial. If a subject cannot independently grant their informed consent in writing, her legal representative may do so in her place.
4. Women of childbearing potential (WOCBP) must perform a pregnancy test at the time of enrollment and agree to the use of a medically acceptable contraceptive method during the selection period and while receiving the medication specified in the protocol. A woman of childbearing age is considered to be any woman physiologically capable of becoming pregnant, from menarche to becoming postmenopausal, unless she is permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menstruation for 12 months without an alternative medical cause. A high level of follicle stimulating hormone (FSH) in the postmenopausal range can be used to confirm a postmenopausal state in women not using hormonal contraceptives or hormone replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

   Only women of childbearing age who adhere to the contraceptive methods recommended by the Clinical Trial Facilitation Group (CTFG) as highly effective contraceptive methods may participate, that is, with a failure rate of less than 1% per year when used consistently and correct:
   * Combined hormonal contraception (containing estrogen and progestin) associated with inhibition of ovulation (oral, intravaginal or transdermal).
   * Progestin-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
   * Intrauterine device (IUD)
   * Intrauterine Hormone Release System (IUS)
   * Bilateral tubal occlusion
   * Vasectomized partner (provided the partner is the participant's only sexual partner in the WOCBP trial and the vasectomized partner has received a medical evaluation of surgical success)
   * Sexual abstinence (defined as abstaining from sexual intercourse for the entire risk period associated with study treatments)
5. Patients without a medical contraindication for the use of i-mTOR.
6. Immunosuppressive induction rATG.

Exclusion Criteria:

1. Subjects may not have a history of type I hypersensitivity or idiosyncratic reactions to drugs ganciclovir (GCV) or valganciclovir (VGCV).
2. Pregnant women.
3. Breastfeeding women.
4. Subjects may not have any clinically significant disease that could interfere with study evaluations.
5. Participation in another clinical trial promoted by the pharmaceutical industry, in which the promoter already establishes in the protocol what the treatment of CMV should be.
6. Patients with active viral replication of the HCV, HBV and / or HIV viruses.
7. Patients requiring a desensitizing treatment that includes plasma exchange, Campath-1, Rituximab®, Eculizumab® and / or Gammaglobulin.
8. Presence of donor-specific antibodies (DSA).
9. Prior intolerance to study medication (Certican®), prior documented history of hereditary galactose intolerance, Lapp's lactase deficiency, or glucose or galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who require initiation of anti-viral treatment with valganciclovir | 3 months
  Proportion of patients who require initiation of anti-viral treatment with valganciclovir after reaching a viral replication threshold greater than 5000IU / ml evaluated in plasma being asymptomatic, comparing the different arms

SECONDARY OUTCOMES:
Incidence of CMV disease | 3 months
  Number of patients with symptomatic CMV disease in each arm
Recurrence of CMV infection after initiation of anti-viral treatment | 3 months
  Number of patients with CMV infection after initiation of anti-viral treatment
Recurrence of CMV infection after switch to everolimus treatment | 3 months
  Number of patients with CMV infection after switch to everolimus treatment
Kinetic of the CMV-specific cellular response | 3 months
  Changes in the CMV-specific cellular response against 2 major CMV antigens (Ie-1 and Pp65) by IFN-γ ELISPOT technique
Titration of anti-CMV antibodies in serum | 3 months
  Changes in the titration of anti-CMV antibodies in serum by ELISA technique
Evaluation of the anti-CMV specific memory B cell response | 3 months
  Changes in CMV-specific memory B cell response by ELISPOT technique
Incidence of acute clinical graft rejection | 3 months
  Number of patients with acute clinical graft rejection
Incidence of acute subclinical graft rejection | 3 months
  Incidence of acute subclinical graft rejection between both study groups evaluated in protocol biopsies 3 months after transplantation
Estimated Glomerular Filtration Rate (eGFR) | 3 months
  Changes in eGFR between both study groups
Incidence of toxic side effects associated with the drug everolimus | 3 months
  Number of toxic side effects associated with the drug everolimus reported
Withdrawal of Everolimus treatment due to Adverse Events | 3 months
  Number of patients that discontinue Everolimus treatment due to Everolimus related Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain